CLINICAL TRIAL: NCT02609802
Title: The Different Analgesic Potency of Sevoflurane and Desflurane at Equi-minimum Alveolar Concentration
Brief Title: The Different Analgesic Potency of Volatile Anesthetics at Equi-MAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Kyoungho Ryu, Clinical assistant professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-09-028
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Orthopedic Disorders
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Anesthesia was maintained with sevoflurane.
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia was maintained with desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia was maintained with sevoflurane in patients undergoing arthroscopic shoulder surgery under general anesthesia and interscalene brachial plexus block.
  Other Names: SEVO
  Arms: Sevoflurane
Drug: Desflurane — Anesthesia was maintained with desflurane in patients undergoing arthroscopic shoulder surgery under general anesthesia and interscalene brachial plexus block.
  Other Names: DES
  Arms: Desflurane

SUMMARY:
The aim of this clinical trial is to evaluate the difference of analgesic potency of sevoflurane and desflurane at equi-minimum alveolar concentration using a surgical pleth index.

DETAILED DESCRIPTION:
Volatile anesthetics vary in their relative hypnotic potencies. Recent studies demonstrated that equi-minimum alveolar concentration of various volatile anesthetics produced different EEG-derived indices such as bispectral index. However, there was no controlled study that demonstrates the difference of analgesic potency. The aim of this clinical trial is to evaluate the difference of analgesic potency of sevoflurane and desflurane at equi-minimum alveolar concentration using a surgical pleth index.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing arthroscopic shoulder surgery
* patients with american society of anesthesiologist physical status I, II
* patients aged 19-65 years
* patients obtaining written informed consent

Exclusion Criteria:

* patients with a history of any psychiatric or neurological disease
* patients who had received any medication affecting the central nervous system
* patients who had received medication affecting the sympathetic or parasympathetic nervous systems
* patients who have not received interscalene approach brachial plexus block (refusal or failure)
* pregnant women

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Analgesic potency of volatile anesthetics | the first 60 min of maintaining a steady state 1 MAC of volatile agents
  The analgesic potency was evaluated by surgical pleth index value

CONTACTS AND LOCATIONS:
Overall Officials: Kyoungho Ryu, M.D., Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided